CLINICAL TRIAL: NCT06148285
Title: Hyperbaric Oxygen Therapy in Acute Ischemic Stroke Recovery
Brief Title: Hyperbaric Oxygen Therapy in Acute Ischemic Stroke Ischemic Stroke Recovery (Pro00061930)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LCMC Health (Other)
Responsible Party: Principal Investigator, Sheryl Martin-Schild, Medical Director of Neurology & Stroke, LCMC Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00061930.1
Record Dates: First submitted 2023-07-22; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- 100% oxygen under 2.0ATA (Experimental): The first intervention arm consists of ischemic stroke patients who would undergo HBOT at 2.0 ATA with 100% oxygenation for 60 minutes x10 treatments (Monday-Friday of two sequential weeks).
  Interventions: Device: Hyperbaric Oxygen Therapy
- 21% oxygen under 2.0ATA (Active Comparator): The second intervention arm would consist of ischemic stroke patients undergoing HBOT at 2.0 ATA with 21% oxygen (room air) for 60 minutes x10 treatments (Monday-Friday of two sequential weeks).
  Interventions: Device: Hyperbaric Oxygen Therapy
- 21% oxygen under 1.14ATA (Sham Comparator): For sham-control; ischemic stroke patients will undergo placement in the hyperbaric oxygen chamber for the same duration of time (60 minutes x10 treatments, Monday-Friday of two sequential weeks) and pressure maintained at 1.14 ATA with 21% oxygen (room air), a non-therapeutic dose of HBOT that sufficiently increases pressure to simulate ear popping, hence maintaining participants blinded to the intervention / sham.
  Interventions: Device: Hyperbaric Oxygen Therapy

INTERVENTIONS:
Device: Hyperbaric Oxygen Therapy — Hyperbaric Oxygen Therapy

SUMMARY:
This study will critically examine the feasibility, safety and efficacy of HBOT during inpatient rehabilitation (IPR) after acute ischemic stroke measured by non-disruption of 3 hours of daily therapy, frequency of neurological deterioration or complications (seizure, hemorrhage, brain edema), and functional communication, activities of daily living (ADLs) and mobility.

DETAILED DESCRIPTION:
Preclinical studies support that HBOT augments several adaptive mechanisms following ischemic stroke, including neuroplasticity, cerebral angiogenesis, and regeneration of nerve fibers. The earlier the treatment, the greater potential for a therapeutic effect. However, logistical issues and safety concerns have prevented application of HBOT in the hyperacute window, particularly when coupled with recanalization therapy as the risk of hemorrhagic conversion is highest, monitoring intervals are short, and the natural history is being altered by another treatment. By enrolling patients who are in the subacute phase of stroke who are admitted to an inpatient rehab facility, the risk of HBOT is lower, monitoring intervals are longer, and the selected population has newly acquired and targetable stroke-related disability. Further, the patients are in a supervised setting and available for daily one-hour treatments without disrupting their intensive multidisciplinary rehab plan thereby minimizing nonadherence to daily treatments. Neuroimaging supports that injured, but not dead, brain cells can persist for months after an ischemic event. Hypoxia mediates cellular activity and death through multiple mechanisms. Ongoing decrease in oxygenation to the damaged area due to impaired blood flow works against cellular repair, recovery, and development of new synaptic connections. Increasing oxygen availability has been considered as an obvious treatment for stroke. HBOT has the potential to facilitate the recovery of injured or inactive neurons through increased blood flow and oxygen delivery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and above
* Ischemic stroke proven on neuroimaging
* Within 7-30 days post-stroke on day 1 of treatment
* Admitted to Touro Inpatient Rehab Facility

Exclusion Criteria:

* Pre-stroke modified Rankin Scale Score >2
* Parenchymal hemorrhagic transformation (PH1 or PH2)
* Receptive aphasia such that recommendations for preventative measures to mitigate barotrauma cannot be followed
* History of recurrent and unprovoked seizures requiring a change in management in the last 3 months to control seizures
* Pulmonary disease requiring supplemental oxygen or daily respiratory medication management (metered dose inhalers, nebulized treatment or steroids)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-05-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy outcome; change in total and subcomponents of functional independence measure (FIM) | 2 weeks
  Difference in the total, motor, and cognitive functional independence measure (FIM) scores between the three arms at the end of respective treatment blocks (2 - week period). Additional analyses for change in the FIM score will also be conducted.
Feasibility outcome; proportion of patients who complete HBOT sessions | 2 weeks
  At least 80% of enrolled patients will be able complete all planned HBOT sessions. HBOT will not directly influence a reduction in quantity or quality of prescribed standard of care rehabilitative therapy.
Safety outcome 1; ear pain | 2 weeks
  Mild to moderate ear pain: absolute difference (AD) vs. control group ≤ 20%.
Safety outcome 2; barotrauma | 2 weeks
  Barotrauma as diagnosed by clinical exam: AD vs. control group ≤ 10%.
Safety outcome 3; any other serious adverse event | 2 weeks
  any of the following absolute difference (AD) vs. control group ≤ 20%: neurological worsening (increase in NIHSS at least 4 points), symptomatic intracranial hemorrhage (parenchymal hemorrhage with neurological worsening), status epilepticus, pulmonary dysfunction (Defined as: respiratory sx requiring supplemental O2, breathing treatment, or evident of pneumothorax or pneumonia on chest imaging performed to evaluate respiratory sx), or death attributed to intervention.

SECONDARY OUTCOMES:
Per-protocol analysis; change in total and subcomponents of functional independence | 2 weeks
  Per-protocol analysis comparing total and sub-component FIM scores among HBOT treated and non-HBOT treated patients who completed all HBOT treatment as per the study protocol.
  Comparison of FIM sub-scores on the FIM functional and cognitive sub-scales. Adjusted estimates of effect of HBOT treatment after controlling for stroke severity (NIHSS), age, pre-morbid mRS evaluated via generalized linear modeling Sub-group analyses for age, sex, race, stroke severity (NIHSS), stroke etiology (TOAST criteria), cortical vs. sub-cortical strokes, pre-morbid disability (pre-morbid mRS)
Adjusted HBOT treatment effect | 2 weeks
  Adjusted estimates of effect of HBOT treatment after controlling for stroke severity (NIHSS), age, pre-morbid mRS evaluated via generalized linear modeling
Sub group analyses to evaluate heterogeneity of treatment effect | 2 weeks
  Sub-group analyses for age, sex, race, stroke severity (NIHSS), stroke etiology (TOAST criteria), cortical vs. sub-cortical strokes, pre-morbid disability (pre-morbid mRS)
Long-term outcome; 90-day good functional outcome vs. significant to severe disability or death | 90 days
  We will compare the proportions of HBOT and non-HBOT treated patients who achieve a 90-day mRS of 0 - 2 (good functional outcome) vs. 3 - 6 (Significant to severe disability or death - SSD) based on intent to treat populations. Additional analyses for the 90-day mRS would include Per-protocol analysis comparing 90-day mRS among HBOT treated and non-HBOT treated patients who completed all HBOT treatments as per the study protocol.
Long-term outcome; 90-day functional outcome evaluated as ordinal shift in the modified Rankin Scale | 90 days
  Ordinal shift in 90-Day mRS across the full scale of mRS for HBOT treated patients vs. non-HBOT treated patients - based on intent to treat and per protocol populations.
Long-term outcome; Adjusted 90-day good functional outcome vs. significant to severe disability or death | 90 days
  Adjusted estimates of effect of HBOT treatment after controlling for stroke severity (NIHSS), age, pre-morbid mRS evaluated via logistic regression - based on intent to treat and per protocol populations.
Long-term outcome; Adjusted 90-day functional outcome evaluated as ordinal shirt in the modified Rankin Scale | 90 days
  Adjusted estimates of effect of HBOT treatment after controlling for stroke severity (NIHSS), age, pre-morbid mRS evaluated via ordinal regression models for proportional differences between treated and non-treated patients - based on intent to treat and per protocol populations.
Long-term outcome; Sub group analyses to evaluate heterogeneity of treatment effect for 90-day outcome | 90 days
  Sub-group analyses for age, sex, race, stroke severity (NIHSS), stroke etiology (TOAST criteria), cortical vs. sub-cortical strokes, pre-morbid disability (pre-morbid mRS)

CONTACTS AND LOCATIONS:
Locations (1):
- Touro Infirmary New Orleans, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Data requests may be submitted 12 months after publication of all planned manuscripts. Data will be made accessible for up to 12 months. Extensions may be considered on a case-by-case basis. Only fully de-identified data elements will be shared with qualified investigators, for use of personal (non-commercial) research. Data will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: Data requests may be submitted 12 months after publication of all planned manuscripts. Data will be made accessible for up to 12 months. Extensions may be considered on a case-by-case basis.
Access Criteria: Only fully de-identified data elements will be shared with qualified investigators, for use of personal (non-commercial) research. Data will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).